CLINICAL TRIAL: NCT03881046
Title: Multidimensional Evaluation Of Daily Living Activities And Quality Of Life In Lung Cancer
Brief Title: Multidimensional Evaluation Of Daily Living Activities And Quality Of Life In Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Hamide Sahin, Multidimensional Evaluation Of Daily Living Activities And Quality Of Life In Lung Cancer Patients, Hacettepe University
Other Study IDs: GO 18/737-08
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lung cancer
- healthy control group

SUMMARY:
The aim of our study was to compare the daily living activities with a performance-based protocol in lung cancer patients and healthy controls.

DETAILED DESCRIPTION:
Lung cancer is the abnormal proliferation of cells in the lung tissue and a mass in the lung. The primary symptoms of this health problem include cough, dyspnea, chest pain, hemoptysis and sputum. In addition to these symptoms, muscle strength, respiratory function and effort level are decreased.

Inadequate daily living activities in cancer patients are expressed.But studies evaluating the activities of daily living in patients with lung cancer are inadequate and patients are evaluated only using scales. For the measurement of functional status in daily living activities, these scales provide important information about the detection of symptoms and the progression of the disease. However, it is very difficult to determine the limitation of perceived difficulty in daily living activities with these scales. In addition, since these scales are a method of measurement, the objectivity is open to discussion. It is thought that a performance-based protocol will facilitate the detection of limitations and provide more objective findings. We think that the Londrina protocol fully reflects the activities of daily living and thus will give us an objective measurement.

This study will show us the problem and its cause in daily life activities in patients with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* To have a diagnosis of lung cancer
* Complete chemotherapy
* Complete radiotherapy
* Coopere,
* Accepts participation in the study will be included in the study

Exclusion Criteria:

* Neurological, cognitive or orthopedic diseases that affect the measurements
* Acute infection
* Individuals with other chronic diseases that may affect their walking will not be included in the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who are diagnosed with Lung Cancer at Hacettepe University and who reffered to the Cardiopulmonary Rehabilitation Unit for Physiotherapy also who are willing to participate in the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Activities Of Daily Living | 1st day
  Daily Living Activities will be evaluated using the Londrina Protocol.The protocol consists of 5 stations. Stations are including organizing books on the table, 18 meters walking by carrying 10% of body weight symmetrically, arranging books by putting them on shelves, hanging the laundry in the laundry basket and walking 18 meters. İndividual will do these activities at his own pace and the time will be recorded at the end.

SECONDARY OUTCOMES:
Life Quality | 1st Day
  Quality of life will be measured using Core Quality of Life Questionnaire (EORTC QLQ-C30) The questionnaire consists of 30 questions and provides information on quality of life and symptoms.
Peripheral Muscle Strength | 1st Day
  Muscle strength will be evaluated by force measuring dynamometer device 3 times. M.Quadriceps Femoris, shoulder abduction, shoulder flexion, elbow flexion, elbow extension and hand grip strength of all cases will be measured.
Dyspnoea | 1st Day
  Dyspnoea will be evaluated using the Medical Research Council Dyspnoea Scale. The Medical Research Council Dyspnoea Scale has a score of 0-4. İn this scoring system 0 indicates that there is no dyspnoea, whereas 4 indicates that the dyspnoea is too high.
Respiratory Functions | 1st Day
  Respiratory functions will be measured by spirometric measurement. This measurement will give us FEV1 FVC FEV1 / FVC values.
Exercise Capacity | 1st Day
  6 Minute walk test will be used.In the test, the person will be asked to walk as fast as possible in a 30-meter corridor and the walking distance will be recorded in 6 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamide Sahin, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes